CLINICAL TRIAL: NCT06081920
Title: A Phase II Study to Evaluate the Safety, Tolerability, and Efficacy of IBI363 in Subjects With Advanced Melanoma
Brief Title: A Study of IBI363 in Subjects With Advanced Melanoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Innovent Biologics (Suzhou) Co. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CIBI363A201
Record Dates: First submitted 2023-10-07; First posted 2023-10-13 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2025-05

CONDITIONS: Melanoma
MeSH Terms: conditions — Melanoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- IBI363 (Experimental)
  Interventions: Biological: IBI363

INTERVENTIONS:
Biological: IBI363 — IBI363 monotherapy

SUMMARY:
This is an open-lable, multicenter Phase II study to evaluate the safety, tolerability, and efficacy of IBI363 in advanced melanoma patients

ELIGIBILITY:
Inclusion Criteria:

1. Histologically and/or cytologically confirmed, unresectable, locally advanced or metastatic melanoma (according to the American Joint Committee on Cancer (AJCC) 8th edition staging III-IV). Progression or recurrence after at least first-line systemic standard treatment.
2. At least one measurable lesion (target lesion) per RECIST v1.1.
3. Eastern Cooperative Oncology Group Performance Status (ECOG PS) of 0 or 1.
4. Life expectancy of 3 months or more.
5. Female subjects of childbearing age or male subjects whose partners are female subjects of childbearing age agree to strictly adopt effective contraceptive measures throughout the entire treatment period and 6 months after the treatment period.

Exclusion Criteria:

1. Pregnant or lactating subjects, or subjects who plan to conceive before, during, or within 6 months after the last dose of the study drug.
2. Active or symptomatic central nervous system metastasis.
3. At baseline (within 7 days before the first administration of the study drug), there were any hematological abnormalities as follows: hemoglobin<90 g/L; Absolute neutrophil count (ANC)<1.5 × 109/L; Platelet count<100 × 109/L.
4. At baseline (within 7 days prior to first administration), there were any serum biochemical abnormalities as follows: Total bilirubin>1.5 × ULN; AST or ALT>3 × ULN; If it is tumor liver metastasis, AST or ALT>5.0 × ULN; Serum creatinine>1.5 × ULN or CCr<45 mL/min, using the Cockcroft Fault formula to calculate CCr (using actual body weight); Albumin<30 g/L.
5. At baseline (within 7 days before first administration), there were any coagulation parameter abnormalities as follows: INR>1.5 × ULN (>3 if receiving anticoagulant therapy with stabilizer dosage) × ULN); PTT (or activated partial thromboplastin time (aPTT))>1.5 × ULN (>3 if receiving anticoagulant therapy with stabilizer dosage) × ULN).
6. History of active thrombosis, deep vein thrombosis, or pulmonary embolism within 4 weeks prior to the first administration of the investigational drug, unless sufficient treatment has been given and the investigator believes that the condition is stable.
7. Uncontrolled bleeding or known tendency to bleed.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2023-10-19 (Actual); Primary Completion 2025-06-06 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
AE（Adverse event） | 2 years
ORR（Objective response rate） | 2 years
DoR（duration of response） | 2 years
PFS (progression free survival) | 2 years
DCR (disease control rate) | 2 years
TTR (time to response) | 2 years
TTP (time to progression) | 2 years

SECONDARY OUTCOMES:
OS（overall survival） | 2 years
PK concentration: IBI363 serum concentration | 2 years
ADA (Anti-drug antibody) | 2 years
Nab (Neutralizing antibody) | 2 years

CONTACTS AND LOCATIONS:
Locations (12):
- China (12):
  - Beijing Cancer Hospital, Beijing, Beijing Municipality
  - Peking University Cancer Hospital & Institute, Beijing, China,, Beijing, Beijing Municipality
  - Fujian Cancer Hospital, Fuzhou, Fujian
  - The Third people's hospital of Zhengzhou, Zhengzhou, Henan
  - Hunan Cancer Hospital, Changsha, Hunan
  - Nanjing Drum Tower Hospital, Nanjing, Jiangsu
  - The first affiliated hospital of Nanchang university, Nanchang, Jiangxi
  - Jilin Cancer Hospital, Changchun, Jilin
  - The first hospital of Jilin University, Changchun, Jilin
  - Qilu Hospital of Shandong university, Jinan, Shandong
  - Shanxi Bethune Hospital, Taiyuan, Shanxi
  - Yunan Cancer Hospital, Kunming, Yunan

IPD SHARING:
Plan to Share IPD: No